CLINICAL TRIAL: NCT04248439
Title: A Phase 2 Clinical Trial to Evaluate the Efficacy of the Infusion of Autologous CD34+ Cells Transduced With a Lentiviral Vector Carrying the FANCA Gene in Pediatric Subjects With Fanconi Anemia Subtype A
Brief Title: Gene Therapy for Fanconi Anemia, Complementation Group A
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP-L102-0319
Record Dates: First submitted 2020-01-24; First posted 2020-01-30 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Fanconi Anemia Complementation Group A
Keywords: anemia; bone marrow failure; gene therapy
MeSH Terms: conditions — Fanconi Syndrome; Anemia; Bone Marrow Failure Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RP-L102 (Experimental): RP-L102 is CD34+ enriched cells from subjects with Fanconi anemia subtype A transduced ex vivo with a lentiviral vector carrying the FANCA gene
  Interventions: Biological: RP-L102

INTERVENTIONS:
Biological: RP-L102 — CD34+ enriched cells from subjects with Fanconi anemia subtype A transduced ex vivo with a lentiviral vector carrying the FANCA gene

SUMMARY:
The objective of this study is to assess the therapeutic efficacy of a hematopoietic cell-based gene therapy for patients with Fanconi anemia, subtype A (FA-A).

Hematopoietic stem cells from mobilized peripheral blood of patients with FA-A will be transduced ex vivo (outside the body) with a lentiviral vector carrying the FANCA gene. After transduction, the corrected stem cells will be infused intravenously back to the patient with the goal of preventing bone marrow failure.

DETAILED DESCRIPTION:
This is a pediatric open-label Phase II clinical trial to assess the efficacy of a hematopoietic gene therapy consisting of autologous CD34+ enriched cells transduced with a lentiviral vector carrying the FANCA gene in subjects with FA-A.

Enriched CD34+ hematopoietic stem cells will be transduced ex vivo with the therapeutic lentiviral vector and infused via intravenous infusion following transduction without any prior conditioning.

ELIGIBILITY:
Inclusion Criteria:

1. Fanconi anemia as diagnosed by chromosomal fragility assay of cultured lymphocytes in the presence of DEB or a similar DNA-crosslinking agent
2. Subject of the complementation group FA-A
3. Minimum age: 1 year and a minimum weight of 8 kg
4. At least 30 CD34+ cells/μL are determined in one bone marrow (BM) aspiration within 3 months prior to CD34+ cell collection OR

6. Provide informed consent in accordance with current legislation 7. Women of childbearing age must have a negative urine pregnancy test at the baseline visit, and accept the use of an effective contraception method during participation in the trial

Exclusion Criteria:

1. Subjects with an available and medically eligible HLA-identical sibling donor.
2. Evidence of myelodysplastic syndrome or leukemia, or cytogenetic abnormalities other than those reported as variant(s) of normal in BM aspirate analysis. This assessment should be made by valid studies conducted within the 3 months before the subject commences the stem cell mobilization/collection procedures of the clinical trial.
3. Subjects with somatic mosaicism associated with stable or improved counts in all PB cell lineages. (If T-lymphocyte chromosomal fragility analysis indicates potential mosaicism, a medically significant decrease (≥1 NCI CTCAE grade) in at least one blood lineage over time must be documented to enable eligibility, as should <5% resistance of bone marrow colony forming cells (CFCs) to 10nM MMC; whenever possible potential mosaicism should also be evaluated by gene sequencing of MMC-resistant CFCs).
4. Lansky performance status ≤60%.
5. Any concomitant disease or condition that, in the opinion of the Principal Investigator, renders the subject unfit to participate in the study.
6. Pre-existing sensory or motor impairment ≥grade 2 according to the criteria of the NCI.
7. Pregnant or breastfeeding women.
8. Hepatic dysfunction as defined by either:

   * Bilirubin >3.0 × the upper limit of normal (ULN) or
   * Alanine aminotransferase (ALT) > 5.0 × ULN or
   * Aspartate aminotransferase (AST) > 5.0 × ULN

   For subjects with bilirubin, ALT or AST above ULN, a workup to identify the etiology of liver abnormality should be conducted prior to confirmation of eligibility as stipulated in exclusion criterion 5, including evaluation of viral hepatitis, iron overload, drug injury or other causes.
9. Renal dysfunction requiring either hemodialysis or peritoneal dialysis.
10. Pulmonary dysfunction as defined by either:

    * Need for supplemental oxygen during the prior 2 weeks in absence of acute infection or
    * Oxygen saturation by pulse oximetry <90%.
11. Evidence of active metastatic or locoregionally advanced malignancy for which survival is anticipated to be less than 3 years.
12. Subject is receiving androgens (i.e. danazol, oxymetholone).
13. Subject is receiving other investigational therapy for treatment/prevention of FA-associated bone marrow failure.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Bone Marrow (BM) Colony-Forming Cell (CFC) Mitomycin-C (MMC) resistance | 21 months
  Bone Marrow (BM) colony-forming cell (CFC) mitomycin-C (MMC) resistance ≥20% at 12 months post-infusion with a confirmatory result at 18 or 21 months (MMC at 10 nM concentration)

SECONDARY OUTCOMES:
Genetic Correction | 24 months
  Evidence of genetic correction as demonstrated by ≥0.1 VCN level of FANCA-LV provirus in total PB cells at 18 months post-infusion with a confirmatory result at 21 or 24 months
Hematologic Stability- Hemoglobin | 24 months
  Hematologic stability demonstrated by hemoglobin levels remaining ≥75% of 6-month post-infusion nadir value, in the absence of Myelodysplastic Syndrome (MDS), Acute Myeloid Leukemia (AML), and/or progressive cytogenetic and/or molecular abnormalities known to be associated with MDS/AML at 18 months post-infusion with a confirmatory result at 21 or 24 months. In settings in which 6-month post-infusion neutrophil or platelet values are demonstrably increased relative to other values during the initial year post-infusion, especially in situations of documented infections or febrile episodes, the value from the most proximate prior visit at which there is no documented infection or febrile episode is used.
  Levels must exceed the following values at the latest documented assessment (≥18 months post-infusion): hemoglobin ≥8 g/dL (National Cancer Institute-Common Terminology Criteria Adverse Events (NCI-CTCAE) v5 Grade <3).
Hematologic Stability- Neutrophils | 24 months
  Hematologic stability demonstrated by neutrophil count remaining ≥75% of 6-month post-infusion nadir value, in the absence of Myelodysplastic Syndrome (MDS), Acute Myeloid Leukemia (AML), and/or progressive cytogenetic and/or molecular abnormalities known to be associated with MDS/AML at 18 months post-infusion with a confirmatory result at 21 or 24 months. In settings in which 6-month post-infusion neutrophil or platelet values are demonstrably increased relative to other values during the initial year post-infusion, especially in situations of documented infections or febrile episodes, the value from the most proximate prior visit at which there is no documented infection or febrile episode is used.
  Levels must exceed the following values at the latest documented assessment (≥18 months post-infusion): neutrophils ≥500/µL (NCI-CTCAE v5 Grade <4).
Hematologic Stability- Platelets | 24 months
  Hematologic stability demonstrated by Platelet count remaining ≥75% of 6-month post-infusion nadir value, in the absence of Myelodysplastic Syndrome (MDS), Acute Myeloid Leukemia (AML), and/or progressive cytogenetic and/or molecular abnormalities known to be associated with MDS/AML at 18 months post-infusion with a confirmatory result at 21 or 24 months. In settings in which 6-month post-infusion neutrophil or platelet values are demonstrably increased relative to other values during the initial year post-infusion, especially in situations of documented infections or febrile episodes, the value from the most proximate prior visit at which there is no documented infection or febrile episode is used.
  Levels must exceed the following values at the latest documented assessment (≥18 months post-infusion): platelets ≥25,000/µL (NCI-CTCAE v5 Grade <4).
Phenotypic Correction | 24 months
  In patients who were not mosaic in Peripheral Blood T-cells prior to gene therapy, the level of phenotypic correction of hematopoietic cells as determined by a T-lymphocyte chromosomal fragility assay targeting a decrease from ≥50% pre-infusion levels to <50% in Peripheral Blood T-cells with DEB-induced aberrations and a ≥20% decrease from pre-treatment levels at ≥182 months post-infusion with a confirmatory result at 21 or 24 months
Safety of RP-L102 | 3 years
  Analysis of Treatment-emergent adverse events (TEAEs), and serious adverse events (SAEs), for the duration of the study.
Tolerability of RP-L102 | 3 years
  Analysis of Treatment-emergent adverse events (TEAEs), and serious adverse events (SAEs), for the duration of the study.
Overall survival | 3 years
  Survival at end of study
Bone Marrow Failure Free Survival | 3 years
  Bone Marrow Failure Free at end of study
Hematological Malignancy Free Survival | 3 years
  Lack of Myelodysplastic Syndrome or Acute Myeloid Leukemia at end of study

CONTACTS AND LOCATIONS:
Overall Officials: Rajni Agarwal, MD, Principal Investigator — Stanford University; Margaret MacMillan, MD, MSc, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of Minnesota, Minneapolis, Minnesota